CLINICAL TRIAL: NCT02727790
Title: Effect of Short Peripheral Electrical Stimulation (PES) on Blood Glucose Lowering Action in Type 2 Diabetes Patients
Brief Title: Effect of Short Peripheral Electrical Stimulation (PES) on Blood Glucose
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 129/12; HTA6446 (Other: Israel: Ministry of Health)
Record Dates: First submitted 2016-02-28; First posted 2016-04-05 (Estimated); Last update posted 2016-06-07 (Estimated); Status verified 2016-03

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Tissue Therapy, Historical

ARMS (2):
- PES Treatment (Experimental): Eligible patients will receive daily 5 min PES treatment for two weeks. Interstitial glucose will be monitored throughout the study using a FreeStyle Navigator (Abbott Diabetes Care, Alameda, CA) continuous glucose monitor (CGM) System
  Interventions: Device: Stimulator
- Control (No Intervention): Interstitial glucose will be monitored throughout the study using a FreeStyle Navigator (Abbott Diabetes Care, Alameda, CA) CGM System

INTERVENTIONS:
Device: Stimulator
  Other Names: BEAC Biomedical Intellistim BE-28TC
  Arms: PES Treatment

SUMMARY:
The epidemic nature of type 2 diabetes mellitus, along with the downsides of current treatments, has raised the need for therapeutic alternatives. The aim of this study is to evaluate safety, tolerability, and the glucose-lowering effect of noninvasive peripheral electrical stimulation (PES) as an alternative treatment for diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with type II diabetes, for at least one year prior to randomization
* Body mass index BMI < 35 Kg/m2
* Stable glucose lowering drugs regimen for at least one month prior to randomization
* Capable of giving informed consent

Exclusion Criteria:

* Pregnancy, or nursing
* 10< HbA1c < 6
* Permanent pacemakers
* Metal prosthesis
* Resting blood pressure > 160/ 100 mmHg
* Skin disease
* Treatment with steroids or beta-blockers treatment with psychiatric medications

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-07; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Number of participants with hypoglycemia, and/ or adverse events that are related to treatment | Baseline through 2 months

SECONDARY OUTCOMES:
Incidence of minor side effects related to treatment | Baseline through 2 months
Changes in mean interstitial glucose levels measured by CGM | Baseline, 1, 2, 5, and 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Assaf-Harofeh Medical Center, Ẕerifin, Israel

REFERENCES:
- [Derived] Catalogna M, Doenyas-Barak K, Sagi R, Abu-Hamad R, Nevo U, Ben-Jacob E, Efrati S. Effect of Peripheral Electrical Stimulation (PES) on Nocturnal Blood Glucose in Type 2 Diabetes: A Randomized Crossover Pilot Study. PLoS One. 2016 Dec 20;11(12):e0168805. doi: 10.1371/journal.pone.0168805. eCollection 2016. PMID 27997608